CLINICAL TRIAL: NCT01212900
Title: The RIGHT Study: Risk Stratification With Image Guidance of HMG Coa Reductase Inhibitor Therapy
Brief Title: Randomized Trial of Imaging Versus Risk Factor-Based Therapy for Plaque Regression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 100214; 10-H-0214
Record Dates: First submitted 2010-09-30; First posted 2010-10-01 (Estimated); Results first posted 2018-10-31 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-02-12

CONDITIONS: Atherosclerosis; Hypercholesterolemia
Keywords: Atherosclerosis; Cardiovascular Disease; Cardiac MRI; Cardiac CT; Cholesterol
MeSH Terms: conditions — Atherosclerosis; Hypercholesterolemia; Cardiovascular Diseases | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Imaging (Experimental): Lipid targets assigned according to the severity of atherosclerotic plaque measured as wall volume in the common and internal carotid arteries by MRI
  Interventions: Drug: Statins, HMG CoA
- Standard (Active Comparator): Standardized statin therapy based on NCEP ATP IIIR guidelines, including clinical risk factors and blood lipid levels.
  Interventions: Drug: Statins, HMG CoA

INTERVENTIONS:
Drug: Statins, HMG CoA — Statin therapy

SUMMARY:
Background:

- Atherosclerosis (thickening of the artery walls caused by cholesterol and other deposits) commonly occurs in the heart vessels and carotid (neck) arteries of adults. This is often present in individuals with high cholesterol levels in their blood. These patients are usually treated with cholesterol lowering medication ( statins ) along with modification of diet and exercise. Researchers are interested in investigating new approaches including magnetic resonance imaging (MRI) and computed tomography (CT) imaging studies to detect blood vessel blockages that would not otherwise be detected by cholesterol levels and risk factors for heart disease.

Objectives:

- To measure atherosclerosis in the heart vessels and carotid arteries using imaging tests (computed tomography (CT) and magnetic resonance imaging (MRI)) before and after standard treatment with cholesterol lowering medication ( statins )

Eligibility:

- Healthy individuals at least 55 years of age who are candidates for therapy to lower their blood cholesterol levels.

Design:

* This study will involve one screening visit and seven study visits over a period of 2 years.
* Participants will be screened with a physical examination and medical history, as well as blood samples and tests to ensure that it is safe for them to have CT and MRI scans. Participants will provide information on current medications, dietary habits, smoking status, alcohol and caffeine intake, and their level of physical activity.
* Participants will be divided into two groups. One group will receive standard doses of medication to lower cholesterol according to current treatment guidelines, while the other group will have MRI scans of the carotid arteries and a CT scan of the heart to determine the best medication dose levels.
* Visits 3 to 5 will be scheduled 3, 6, and 9 months after visit 2. During these visits, researchers will monitor for possible side effects and may change or adjust medications and doses.
* At visit 6, participants will have an MRI scan of the carotid arteries, a physical examination, and blood tests. Medications may be changed or adjusted.
* At visit 7, participants will have blood tests, and medications may be changed or adjusted.
* At the final visit, participants will have MRI and CT scans of the carotid arteries and heart, respectively, as well as a final physical examination and blood tests.

DETAILED DESCRIPTION:
The overall aim of this proposal is to compare the effectiveness of an image guided approach to lipid lowering to standard therapy guided by clinical risk factors and blood lipid levels. Men and women over age 55 who are candidates for statin therapy will be randomized to usual cholesterol lowering care, or to care guided by MRI images of the carotid arteries. Participants randomized to the second, imaging guided, group will be assigned to LDL cholesterol targets according to the degree of atherosclerosis seen by MRI. The study endpoints will be the total degree of plaque regression seen, the dosage of statin drugs required to achieve that reduction, and the rate of cardiovascular events.

FDG-PET is hypothesized to enable visualization of anti-inflammatory effects of statins that most likely occur before anatomic regression of the plaques can be demonstrated on MRI. A pilot substudy is to be conducted to explore this relationship. A subgroup of patients participating in the main study will be asked to participate in FDG PET imaging. The purpose of this pilot study is to determine if FDG avid lesions undergo a greater degree of morphologic regression with therapy controlling for the reduction in LDL cholesterol and the dosage of statins required to achieve that target.

Although contrast-enhanced coronary CT angiography (CTA) with multidetector computed tomography (MDCT) has been used extensively to characterize coronary artery plaque composition, there is little data regarding its reproducibility. A recent study demonstrated excellent reproducibility for this technique but this study was performed using the older 64 detector row CT scanners2. A pilot substudy will be conducted to study the reproducibility of coronary CT angiography using the newer generation of 320 detector row CT scanners.

ELIGIBILITY:
* INCLUSION CRITERIA:

A. Men and Women greater than or equal to 55 years of age

B. Candidates for lipid lowering therapy under NCEP ATP III guidelines without contraindication to statin therapy

C. Willing to modify therapy to enroll in the study

D. Willing to travel to the NIH for follow-up visits.

E. Able to understand and sign informed consent

F. Lab Eligibility parameters:

* eGFR > 45 mL/min/m2
* For age >60 test GFR within 1 week prior to contrast; For age less than or equal to 60 test within 4 weeks

INCLUSION CRITERIA FOR THE PET SUBSTUDY:

Participants who are not participating in the CT Reproducibility study are eligible.

INCLUSION CRITERIA FOR THE REPRODUCIBILITY SUBSTUDY:

Patients will be selected who had a one RR interval initial CT scan with less that 10.5 mSv estimated radiation dosage and who will not be participating in the PET Substudy.

EXCLUSION CRITERIA:

A. Ineligibility for MR imaging due to:

* Previous pacemaker implantation
* Automatic implantable cardioverter-defibrillator (AICD)
* Metal implants or other ferromagnetic devices, or
* Foreign material

B. Claustrophobia

C. Contra-indication or allergy to statin medications.

D. Current statin therapy at or above the maximum dosage permitted per study protocol.

E. Use of fibrates, ezetimibe, niacin, or bile acid binding agents within 6 months of screening visit.

F. Pregnancy and nursing.

G. Liver failure defined clinically and by laboratory data.

H. Mental, neurologic or social condition preventing understanding of the rationale, procedures, risks and potential benefits associated with the trial.

I. Any other conditions that precludes safety for MRI and/or CT imaging per the researcher s evaluation.

EXCLUSION FOR PARTICIPATION FOR GADOLINUIM CONTRAST. PARTICIPANTS MAY STILL UNDERGO ALL OTHER STUDY EVALUATIONS.

(Inclusive of the above exclusion criteria):

1. Allergy to gadolinium for scans using contrast; will be eligible for non-contrast scans.
2. Acute renal failure, renal transplant, dialysis and renal failure (eGFR < 45 mL/min/m2 and/or clinically diagnosed).
3. Individuals with a history of liver transplant or severe liver disease.<TAB>
4. Individuals with hemoglobinopathies or severe asthma.

EXCLUSION FOR PARTICIPATION FOR IODINATED CONTRAST. PARTICIPANTS MAY STILL UNDERGO ALL OTHER SUDY EVALUATIONS.

Prior hypersensitivity reaction to iodinated contrast injection, renal dysfunction (defined as eGFR < 45 mL/min/ m2) or a current clinical diagnosis of renal failure.

EXCLUSION CRITERIA FOR THE PET SUBSTUDY:

Patients who are unable or unwilling to comply with the physical activity restrictions or fast for 12 hours prior to FDG PET scanning will be excluded. Due to the need for dietary manipulation and the maintenance of strict glycemic control we will exclude diabetic patients from our initial study sample. Blood glucose measurements before injection must be within normal limits, less than 200 mg/dL (11 mmol/L).

EXCLUSION CRITERIA FOR THE REPRODUCIBILITY

Patients who did not have a one RR interval initial CT scan. Patients who will participate in the PET Substudy.

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2010-09-30; Primary Completion 2016-11-30 (Actual); Study Completion 2017-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nehal N Mehta, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Zavodni AE, Wasserman BA, McClelland RL, Gomes AS, Folsom AR, Polak JF, Lima JA, Bluemke DA. Carotid artery plaque morphology and composition in relation to incident cardiovascular events: the Multi-Ethnic Study of Atherosclerosis (MESA). Radiology. 2014 May;271(2):381-9. doi: 10.1148/radiol.14131020. Epub 2014 Mar 4. PMID 24592924
- [Background] Polak JF, Szklo M, Kronmal RA, Burke GL, Shea S, Zavodni AE, O'Leary DH. The value of carotid artery plaque and intima-media thickness for incident cardiovascular disease: the multi-ethnic study of atherosclerosis. J Am Heart Assoc. 2013 Apr 8;2(2):e000087. doi: 10.1161/JAHA.113.000087. PMID 23568342
- [Background] Sibley CT, Vavere AL, Gottlieb I, Cox C, Matheson M, Spooner A, Godoy G, Fernandes V, Wasserman BA, Bluemke DA, Lima JA. MRI-measured regression of carotid atherosclerosis induced by statins with and without niacin in a randomised controlled trial: the NIA plaque study. Heart. 2013 Nov;99(22):1675-80. doi: 10.1136/heartjnl-2013-303926. Epub 2013 Jul 19. PMID 23872591
- [Derived] Sandfort V, Lai S, Ahlman MA, Mallek M, Liu S, Sibley CT, Turkbey EB, Lima JA, Bluemke DA. Obesity Is Associated With Progression of Atherosclerosis During Statin Treatment. J Am Heart Assoc. 2016 Jul 13;5(7):e003621. doi: 10.1161/JAHA.116.003621. PMID 27413040
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-H-0214.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Imaging | Standard
Started | 116 | 114
Completed | 104 | 107
Not Completed | 12 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Imaging | Standard | Total
Number analyzed (Participants) | 116 | 114 | 230
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 61 | 51 | 112
  >=65 years | 55 | 63 | 118
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 45 | 92
  Male | 69 | 69 | 138
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 115 | 110 | 225
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 3 | 5 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 11 | 17
  White | 105 | 95 | 200
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean of Wall Volume of Internal Carotid Arteries
Description: Wall volume of internal carotid arteries was measured using magnetic resonance imaging. Participants will undergo 2D and 3D carotid MRI using a 3 Tesla scanner and surface carotid coils. Participants with mild or no atherosclerosis, defined as the lowest tertile of wall volume, will have statin therapy adjusted to a target range of 100-130 mg/dL. Participants in the middle tertile will receive statin therapy adjusted to achieve a target LDL 70-100 mg/dL. Participants with the most severe atherosclerosis will receive statin therapy to an LDL target between 40 and 70 mg/dL. Participants in the Standard arm will have lipid sub-fraction targets determined according to estimated 10 year cardiovascular risk, as per standard NCEP guidelines.
Time Frame: 24 months
Population: The analyses included only those subjects who were assigned standardized statin doses based on imaging of carotids at baseline based on NCEP ATP IIIR guidelines.
Measure: Mean (95% Confidence Interval); unit: Other - mm^3 ( cubic millimeter )
Arm/Group | Imaging | Standard
Number analyzed (Participants) | 91 | 89
Other - mm^3 ( cubic millimeter ) | -3.52 [-7.552305 to 0.506032] | -5.91 [-10.9683601 to -0.8536061]

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Imaging | Standard
All-Cause Mortality (participants affected / at risk) | 0/116 | 1/114
Serious Adverse Events (participants affected / at risk) | 18/116 | 18/114
Other Adverse Events (participants affected / at risk) | 58/116 | 51/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imaging (N=116) | Standard (N=114)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Blood creatine abnormal (Investigations) | 1 | 0
Haemoglobin abnormal (Investigations) | 1 | 0
Hepatic enzyme abnormal (Investigations) | 1 | 3
Hospitalisation (Investigations) | 0 | 1
adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Biopsy skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gingival cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Spinal cord herniation (Nervous system disorders) | 1 | 0
Amnesia (Psychiatric disorders) | 1 | 0
Epiglottitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aortic surgery (Surgical and medical procedures) | 1 | 0
Arthroscopic surgery (Surgical and medical procedures) | 3 | 3
Breast conserving surgery (Surgical and medical procedures) | 0 | 1
Cardiac ablation (Surgical and medical procedures) | 1 | 0
Coronary arterial stent insertion (Surgical and medical procedures) | 0 | 1
Elective procedure (Surgical and medical procedures) | 1 | 0
Hospitalisation (Surgical and medical procedures) | 0 | 1
Prostatectomy (Surgical and medical procedures) | 0 | 1
Thyroidectomy (Surgical and medical procedures) | 1 | 0
Transurethral prostatectomy (Surgical and medical procedures) | 0 | 1
Uterine prolapse repair (Surgical and medical procedures) | 0 | 1
Carotid artery aneurysm (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imaging (N=116) | Standard (N=114)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Hyperbilirubinaemia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Chest discomfort (Cardiac disorders) | 0 | 1
Dyspnoea (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 2 | 1
Presyncope (Cardiac disorders) | 1 | 0
External ear pain (Ear and labyrinth disorders) | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Otitis externa (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Goitre (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 0
Retinal haemorrhage (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 1
Glossodynia (Gastrointestinal disorders) | 1 | 0
nausea (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 2 | 0
fatigue (General disorders) | 3 | 3
Nodule (General disorders) | 0 | 2
Oedema (General disorders) | 2 | 0
Haemangioma of liver (Hepatobiliary disorders) | 0 | 1
Genitourinary tract infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Spinal cord herniation (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Blood creatine abnormal (Investigations) | 0 | 2
Blood pressure increased (Investigations) | 1 | 3
Intraocular pressure increased (Investigations) | 0 | 1
Low density lipoprotein increased (Investigations) | 0 | 1
Pregnancy test false positive (Investigations) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Oedema peripheral (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Fracture (Musculoskeletal and connective tissue disorders) | 2 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle contractions involuntary (Musculoskeletal and connective tissue disorders) | 3 | 0
Muscle rupture (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1
myalgia (Musculoskeletal and connective tissue disorders) | 3 | 5
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Rotator cuff repair (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Upper limb fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 1
Facial paralysis (Nervous system disorders) | 1 | 0
Facial spasm (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 3
Parkinson's disease (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Trigeminal neuralgia (Nervous system disorders) | 0 | 1
Amnesia (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Flank pain (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Urinary tract infection (Renal and urinary disorders) | 0 | 1
Adductor vocal cord weakness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Adenoviral upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chest discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
Acupuncture (Surgical and medical procedures) | 1 | 0
Antidepressant therapy (Surgical and medical procedures) | 1 | 0
Breast operation (Surgical and medical procedures) | 1 | 0
Cyst drainage (Surgical and medical procedures) | 0 | 1
Finger amputation (Surgical and medical procedures) | 0 | 1
Hernia repair (Surgical and medical procedures) | 1 | 0
Meniscus operation (Surgical and medical procedures) | 1 | 0
Radioactive iodine therapy (Surgical and medical procedures) | 0 | 1
Rotator cuff repair (Surgical and medical procedures) | 1 | 0
Tendon operation (Surgical and medical procedures) | 1 | 0
Vocal cord polypectomy (Surgical and medical procedures) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Intermittent claudication (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/00/NCT01212900/Prot_SAP_000.pdf